CLINICAL TRIAL: NCT02492048
Title: Effectiveness of CelluTome Epidermal Harvesting System in Autologous Skin Grafting of Chronic Wound Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: LifeBridge Health (Other)
Collaborators: Kinetic Concepts, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2199
Record Dates: First submitted 2015-07-01; First posted 2015-07-08 (Estimated); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Wounds and Injuries
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Split Thickness Skin Graft Harvest (Active Comparator): Retrospective review
  Interventions: Procedure: Split Thickness Skin Graft
- Cellutome Epidermal Harvesting System (Experimental): Prospective patients will receive a skin graft utilizing the Cellutome Epidermal Harvesting System
  Interventions: Device: Cellutome Epidermal Harvesting System

INTERVENTIONS:
Device: Cellutome Epidermal Harvesting System — Cellutome Epidermal Harvesting System
  Arms: Cellutome Epidermal Harvesting System
Procedure: Split Thickness Skin Graft — Split Thickness Skin Graft
  Arms: Split Thickness Skin Graft Harvest

SUMMARY:
This is multi-center prospective, longitudinal case series with comparison to historical controls.

DETAILED DESCRIPTION:
The primary objective to this study is to determine the effectiveness of CelluTome™ epidermal harvesting system as an outpatient skin grafting system for selected patients versus inpatient skin graft harvest. This is multi-center prospective, longitudinal case series with comparison to historical controls. In this study, all subjects will receive the same treatment protocol regardless of institution. This will include routine wound photography. Ongoing healing process will be recorded and reviewed. The secondary objectives of this study are to establish an ideal donor site size, recipient site size and ideal patient population (especially high operative risk patients) that would benefit from the use of CelluTome™ Epidermal Harvesting System.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* Patients requiring split-thickness skin grafting with non-infected wounds
* Age of participants: 18 years and above at the time of informed consent
* Gender: Male or Female
* Subjects who will be locally available for the next 6 months.

Exclusion Criteria:

* Infected chronic wound
* Patients who are unable to adhere to scheduled study visits
* Patients who have severe arterial insufficiency requiring vascular intervention to restore adequate blood flow
* Patients who have an active drug/alcohol dependence or abuse history
* Use of Investigational Agents/Devices on study or within 30 days prior to informed consent or within 30 days prior to use of device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-12-16 (Actual); Primary Completion 2016-11-22 (Actual); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Healing Time | 8 weeks
  Healing time is defined as the required time for the graft site to become dry enough for removal of the dressing without further discharge from the wound AND 100% re-epithelialization has occurred

SECONDARY OUTCOMES:
Healing at Donor Site | 8 weeks
  Photography and physician examination with determination
Scarring | 8 weeks
  Areas of donor site which heal with excess scar tissue and recipient site which heal due to secondary intention (epithelization without skin grafting application). Photography and physician examination with determination.
Complications | 8 weeks
  Cellulitis involving the donor or recipient site, infection involving continuous drainage, abscess formation, erythema, edema, pruritus and fever. Physician determination of complications post procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Noman A Siddiqui, DPM, MHA, Principal Investigator — Rubin Institute for Advanced Orthopedics, Sinai Hospital of Baltimore, LifeBridge Health
Locations (1):
- Rubin Institute for Advanced Orthopedics, Sinai Hospital of Baltimore, LifeBridge Health, Baltimore, Maryland, United States